CLINICAL TRIAL: NCT00004939
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of 3,4-Diaminopyridine for Demyelinating Polyneuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Mayo Clinic (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11963; MAYOC-585
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
Keywords: demyelinating neuropathy; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Drug: ,4-diaminopyridine

SUMMARY:
OBJECTIVES:

I. Assess the efficacy of 3,4-diaminopyridine in patients with stable chronic demyelinating polyneuropathy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are randomly assigned to oral 3,4-diaminopyridine (3,4-DAP) or placebo administered for 4 days. After a washout of at least 5 days, patients cross to the alternate therapy for 4 days.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Clinical diagnosis of demyelinating neuropathy, i.e.: Hereditary motor and sensory neuropathy type I Chronic inflammatory demyelinating polyneuropathy meeting American Academy of Neurology AIDS Task Force criteria Multifocal motor neuropathy and conduction block Clinically stable for at least 6 months prior to entry --Prior/Concurrent Therapy-- At least 6 months since change in immunosuppressive dose --Patient Characteristics-- Age: 20 to 80 Hepatic: No predisposition to hepatic disease Renal: No predisposition to renal disease Cardiovascular: No predisposition to cardiac disease Other: No other medical condition affecting neuropathy or study evaluation No predisposition to seizures

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 1996-08; Study Completion 1996-08

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. Windebank, Study Chair — Mayo Clinic

REFERENCES:
- [Background] Russell JW, Windebank AJ, Harper CM Jr. Treatment of stable chronic demyelinating polyneuropathy with 3,4-diaminopyridine. Mayo Clin Proc. 1995 Jun;70(6):532-9. doi: 10.4065/70.6.532. PMID 7776711